CLINICAL TRIAL: NCT06549127
Title: Research on Clinical Safety and Effectiveness of Wearable Assistive Devices With Flexible Structure for Daily Life Support of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2023-0009
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): This group is evaluated on three conditions.
  Interventions: Device: Soft Wearable Robot

INTERVENTIONS:
Device: Soft Wearable Robot — This study aims to enroll 20 participants who will receive assistance in flexion and extension of the knee and hip during overground walking adaptation training. Following the initial assessment, participants will undergo three 30-minute sessions of overground walking adaptation training with a powered hip assistive device over two weeks. After completing these sessions, Post-intervention Assessment 1 will be conducted. Then, participants will undergo three 30-minute sessions of overground walking adaptation training with a powered knee assistive device over two weeks, followed by Post-intervention Assessment 2. Each participant will have a total of nine visits, including three functional assessments and six adaptation training sessions. The first visit will involve scheduling subsequent visits. The familiarization process will occur two to three times per week, adjustable for participants' convenience, with each set of three visits completed within three weeks.

SUMMARY:
Gait independence is a critical goal for stroke patients and significantly impacts their return to society. Due to hemiplegia, stroke patients often face walking difficulties. Compensatory approaches using lower limb assistive devices have shown promise in improving independent walking. Wearable assistive devices, which minimize daily life restrictions, are gaining attention globally. Despite the availability of many imported rehabilitation assistive devices, their high cost and poor fit for East Asian patients highlight the need for domestic alternatives. In light of the global interest in robotics, there is a shortage of domestic research on advanced wearable robots. This study aims to clinically test and verify the effectiveness of a flexible, wearable robotic assistive device developed by Angel Robotics for stroke patients.

DETAILED DESCRIPTION:
The study will enroll 20 participants, providing knee and hip assistance during overground walking adaptation training. Participants will undergo an initial assessment followed by three 30-minute sessions of training with a powered hip assistive device over two weeks. Post-intervention Assessment 1 will follow this training. Then, participants will undergo three 30-minute sessions of training with a powered knee assistive device over the next two weeks, followed by Post-intervention Assessment 2. Each participant will have nine visits in total, including three functional assessments and six adaptation training sessions. The schedule for subsequent visits will be arranged during the first visit. The familiarization process will be conducted two to three times per week, adjusted for participants' convenience, with each set of three visits completed within three weeks. Trained therapists will handle the attachment and adjustment of the powered assistive devices.

Assessments will be conducted at three points: before the first training session, after the third session, and after the sixth session. Measurements will be taken under three conditions: without the assistive device, with the assistive device but without power assistance, and with the assistive device and power assistance, in random order.

This study will evaluate the following: Gait speed using the 10-meter walk test, Walking distance using the 6-minute walk test, 3D gait analysis (Human body model) assessing kinetics and kinematics, Energy consumption, including oxygen rate (VO2/ml/min per kg of body weight) and oxygen cost (oxygen rate per walking speed in m/min), Lower limb strength and motor function, assessed by the Functional Ambulatory Category (gait independence), Berg Balance Test (balance ability), and Rivermead Mobility Index (motor ability), These evaluations will help determine the effectiveness of the wearable robotic assistive device in aiding the gait of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients aged 19 years and older 2. Diagnosed with stroke confirmed by neurologists or neurosurgeons through imaging techniques such as CT or MRI 3. Chronic hemiplegic stroke patients, 6 months or more post-stroke onset 4. Patients with a Functional Ambulatory Category (FAC) score of 3 or higher 5. Patients with a Mini-Mental State Examination (MMSE) score of 10 or higher, who can understand the study, have a voluntary willingness to participate, and have given consent to participate

Exclusion Criteria:

* 1. Acute/subacute stroke patients within 6 months of stroke onset 2. Quadriplegia 3. Ataxia 4. Severe lower limb joint contractures that make wearing the assistive device difficult 5. Patients with neurological, musculoskeletal, or cardiopulmonary diseases that affect walking 6. Any other conditions deemed inappropriate for participation in the study by the researcher

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
10-meter walking test | Initial Assessment
  The 10 Meter Walk Test (10MWT) is a simple and commonly used assessment to evaluate walking speed. During the test, participants are instructed to walk a distance of 10 meters. The time is measured for the middle 6 meters, allowing the first and last 2 meters for acceleration and deceleration. This approach ensures a more accurate assessment of the participant's steady-state walking speed.
10-meter walking test | After 2 weeks of hip assistive device adaptation training
  The 10 Meter Walk Test (10MWT) is a simple and commonly used assessment to evaluate walking speed. During the test, participants are instructed to walk a distance of 10 meters. The time is measured for the middle 6 meters, allowing the first and last 2 meters for acceleration and deceleration. This approach ensures a more accurate assessment of the participant's steady-state walking speed.
10-meter walking test | After 2 weeks of knee assistive device adaptation training
  The 10 Meter Walk Test (10MWT) is a simple and commonly used assessment to evaluate walking speed. During the test, participants are instructed to walk a distance of 10 meters. The time is measured for the middle 6 meters, allowing the first and last 2 meters for acceleration and deceleration. This approach ensures a more accurate assessment of the participant's steady-state walking speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No